CLINICAL TRIAL: NCT05407493
Title: Comparison of a Double-layered Technique With the Buccal Sliding Flap for Closure of Oroantral Communication
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Prof, University of Siena
Other Study IDs: ODO002, 26/06/2020
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Oroantral Fistula
MeSH Terms: conditions — Oroantral Fistula

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Buccal flap: The buccal flap is slid over the fistula and sutured to the undermined palatal mucosa using horizontal mattress sutures.
- Double-layer: A combination between a buccal trapezoidal flap and a palatal connective pedicle flap.
- Buccal flap with L-PRF: A L-PRF plug is interposed between the fistula and the buccal sliding flap.

SUMMARY:
The aim of this study is to compare the clinical results of combining a pedicle connective palatal flap with a trapezoid buccal flap with the standard buccal flap alone in the closure of oro-antral fistula (OAF), and the buccal flap combined with leukocyte and platelet rich fibrin.

ELIGIBILITY:
Inclusion Criteria:

Eligible population among those older than 18 y.o, systemically healthy, with a diagnosis of OAC (OroAntral Communication), or with a strong pre-extractive radiographic suspicion of potential OAC, and associated symptoms (varying among cheek pain with nasal obstruction, purulent rhinorrhea, foul odor, foul taste, headaches, anterior maxillary tenderness, and postnasal drip) .

Exclusion Criteria:

i) received antibiotic therapy in the last 3 months ii) requiring anticoagulation therapy iii) had systemic diseases that could interfere with oral tissue healing process/bleeding iv) were using bisphosfonates v) were pregnant vi) had mental/physical disabilities vii) underwent radiation treatment to the head or neck region.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible patients with a clinical diagnosis of oroantral fistula among those referring to the Dental department of Siena University Hospital
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Closure success | One month after surgery
  Measured with probing and Valsalva test

SECONDARY OUTCOMES:
Patient reported Pain | Each week for one month
  Pain on a VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Discepoli, Study Director — University of Siena
Locations (1):
- Dipartimento di Odontostomatologia, Siena, Italy